CLINICAL TRIAL: NCT03040362
Title: A Phase 1 Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-Lasmiditan Following Single Oral Dose Administration in Healthy Male and Female Subjects
Brief Title: Absorption, Metabolism and Excretion of [14C]-Lasmiditan - Single Oral Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: CoLucid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16884; H8H-CD-LAHH (Other: Eli Lilly and Company); COL MIG-110 (Other: CoLucid Pharmaceuticals)
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2018-01

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-lasmiditan (Experimental): [14C]-lasmiditan administered as a 200 mg (approximately 100 µCi) oral solution
  Interventions: Drug: [14C]-lasmiditan

INTERVENTIONS:
Drug: [14C]-lasmiditan — [14C]-lasmiditan as a 200 mg (approximately 100 µCi) oral solution
  Other Names: LY573144

SUMMARY:
This study will be an open-label, nonrandomized, absorption, metabolism, and excretion study of [14C]-lasmiditan administered as a 200-milligrams (mg) (approximately 100 microcuries[µCi]) oral solution to 8 healthy males and females, following at least a 10 hour fast from food to assess the pharmacokinetics (PK), metabolism, and routes and extent of elimination of a single oral dose of 200 mg (approximately 100 µCi) [14C] lasmiditan in healthy males and females.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, between 18 and 60 years of age, inclusive, at Screening
* Have a body mass index range of 18.5 to 32.0 kilograms per meter squared (kg/m²), inclusive, at Screening
* In good health, determined by no clinically significant findings from medical history, 12 lead electrocardiogram (ECG), and vital signs measurements at Screening or Check-in (Day 1) as determined by the Investigator (or designee)
* Clinical laboratory evaluations (including clinical chemistry panel [fasted at least 10 hours], hematology/complete blood count [CBC], and urinalysis [UA]; within the reference range for the test laboratory at Screening and Check-in, unless deemed not clinically significant by the Investigator (or designee)
* Negative test for selected drugs of abuse at Screening (does not include alcohol) and at Check-in (does include alcohol)
* Negative hepatitis panel (including hepatitis B surface antigen and hepatitis C virus antibody and negative human immunodeficiency virus (HIV) antibody screens
* Females must be nonpregnant, nonlactating, and either postmenopausal (defined as no menstrual period for at least 12 months and confirmed by a serum follicle-stimulating hormone (FSH) level of ≥40 milli-international units (mIU/mL), surgically sterile (e.g., bilateral oophorectomy, salpingectomy, and/or hysterectomy) for at least 90 days prior to Screening, or must have undergone bilateral tubal ligation and agree to use effective contraception. For all females, the pregnancy test results must be negative at Screening and Check-in
* Males will be surgically sterile for at least 90 days prior to Screening or when sexually-active with female partners of child-bearing potential will agree to use contraception from Check-in until 90 days following Discharge. Male participants must also be willing to refrain from donating sperm from Check-in until 90 days following Discharge
* Able to comprehend and willing to sign an informed consent form (ICF)
* A minimum of 1 to 2 bowel movements per day

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, infectious, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the Investigator [or designee]) prior to Check-in
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee) prior to Check-in
* History of stomach or intestinal surgery or resection that could alter absorption or excretion of orally administered drugs prior to Check-in, except that cholecystectomy, appendectomy, and hernia repair will be allowed if it was not associated with complications
* History or presence of an abnormal ECG that, in the Investigator's (or designee's) opinion, is clinically significant at Screening or Check-in
* History of orthostatic hypotension with or without syncope
* A sustained seated systolic blood pressure >150 millimeters of mercury (mmHg) or <90 mmHg or a diastolic blood pressure >90 mmHg or <50 mmHg at Screening or Check in. Blood pressure may be retested twice at intervals of 5 minutes. The out of range blood pressure values will be considered sustained if either the systolic or diastolic blood pressures are outside the stated limits after these 3 assessments
* History of alcoholism or drug addiction within 1 year prior to Check-in
* Use of any tobacco- or nicotine-containing products (including but not limited to cigarettes, e-cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to Check-in, or positive cotinine screen at Screening or Check-in
* Participation in more than 1 other radiolabeled investigational study drug trial within 12 months prior to Check-in. The previous radiolabeled study drug must have been received more than 6 months prior to Check-in for this study and the total exposure from this study and the previous study will be within the recommended levels considered safe, per United States (US) Title 21 Code of Federal Regulations (CFR) 361.1 (e.g., less than 5,000 millirem [mrem] whole body annual exposure)
* Exposure to significant radiation (e.g., serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months prior to Check-in
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives (if known) or 30 days prior to Check-in, whichever is longer
* Use of any prescription medications/products within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee)
* Use of any over-the-counter, nonprescription preparations (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days prior to Check-in, unless deemed acceptable by the Investigator (or designee)
* Poor peripheral venous access prior to Check-in
* Donation of whole blood from 56 days prior to Screening through Discharge, inclusive, or of plasma from 30 days prior to Screening through Discharge, inclusive
* Receipt of blood products within 2 months prior to Check-in
* Participant is at imminent risk of suicide (positive response to question 4 or 5 on the baseline Columbia-Suicide Severity Rating Scale (C-SSRS) or had a suicide attempt within 6 months prior to Screening
* Any acute or chronic condition that, in the opinion of the Investigator (or designee), would limit the particpant's ability to complete or participate in this clinical study
* Any other unspecified reason that, in the opinion of the Investigator (or designee) or Sponsor, makes the participant unsuitable for enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-05-06 (Actual); Study Completion 2017-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were preceded by an overnight fast (at least 10 hours) from food (not including water) before receiving a dose of [14C]-lasmiditan.
Groups:
- [14C]-Lasmiditan: Participants were administered a single oral dose of radiolabeled [14C]-lasmiditan as a 200 mg (approximately 100 µCi) oral solution on Day 1.
Period: Overall Study
Arm/Group | [14C]-Lasmiditan
Started | 8
Received at Least 1dose of Study Drug | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Arm/Group | [14C]-Lasmiditan
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed concentration based on plasma concentrations of lasmiditan.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, and 192 hours post-dose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable [14C]-lasmiditan PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | [14C]-Lasmiditan
Number analyzed (Participants) | 8
nanograms per milliliter (ng/mL) | 299 (36)

2. Primary Outcome: Pharmacokinetics: Time of Maximum Observed Plasma Concentration (Tmax)
Description: Time to maximum concentration based on plasma concentrations of lasmiditan.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, and 192 hours pos-tdose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable [14C]-lasmiditan PK data.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | [14C]-Lasmiditan
Number analyzed (Participants) | 8
hours (hr) | 2.02 [2.00 to 3.00]

3. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Tlast (AUC[0-tlast])
Description: Area under concentration time curve (AUC) from Hour 0 to the last measurable concentration based on plasma concentrations of lasmiditan.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, and 192 hours post-dose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable [14C]-lasmiditan PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | [14C]-Lasmiditan
Number analyzed (Participants) | 8
nanogram*hour per milliliter (ng*h/mL) | 2100 (38)

4. Primary Outcome: AUC Time Zero to Infinity (AUC0-∞) Blood/Plasma Ratio
Description: AUC time zero to infinity (0-∞) of total radioactivity in blood/AUC0-∞ of total radioactivity in plasma.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, and 192 hours post-dose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable [14C]-lasmiditan PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | [14C]-Lasmiditan
Number analyzed (Participants) | 8
Ratio | 0.948 (6)

5. Primary Outcome: AUC Time Zero to Infinity (AUC0-∞) Plasma Lasmiditan/Total Radioactivity Ratio
Description: AUC time zero to infinity (0-∞) of lasmiditan in plasma/AUC0-∞ of total radioactivity in plasma.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, and 192 hours pos-tdose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable [14C]-lasmiditan PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | [14C]-Lasmiditan
Number analyzed (Participants) | 8
Ratio | 0.131 (18)

6. Secondary Outcome: Pharmacokinetics - Cumulative Amount of Lasmiditan and Its Metabolites Excreted in Urine
Description: Amount of Lasmiditan and its metabolites (M3, M7, M8, (S,R)-M18, and (S,S)-M18) excreted in urine (Aeu) over sampling interval.
Time Frame: Pre-dose (-12 to 0 hours) and intervals: 0 to 6, 6 to 12, 12 to 24, 24 to 48, 48 to 72, 72 to 96, 96 to 120, 120 to 144, 144 to 168, and 168 to 192 hours post-dose
Population: All enrolled participants who received at least one dose of the study drug and had evaluable [14C]-lasmiditan PK data.
Measure: Mean (Standard Deviation); unit: milligram (mg)
Arm/Group | [14C]-Lasmiditan
Number analyzed (Participants) | 8
milligram (mg)
  Lasmiditan | 5.81 (1.12)
  M3 | 1.62 (0.506)
  M7 | 0.00224 (0.000902)
  M8 | 132 (10.8)
  (S,R)-M18 | 1.85 (0.534)
  (S,S)-M18 | 0.445 (0.127)

7. Secondary Outcome: Percentage of Lasmiditan Recovered in Urine, Relative to Dose Administered
Description: Percentage of lasmiditan recovered in urine (%UR), relative to dose administered calculated as %UR = 100 (amount of lasmiditan excreted in urine over a sampling interval (Aeu)/dose).
Time Frame: as for outcome 6
Population: All enrolled participants who received at least one dose of the study drug and had evaluable [14C]-lasmiditan PK data.
Measure: Mean (Standard Deviation); unit: % of lasmiditan dose
Arm/Group | [14C]-Lasmiditan
Number analyzed (Participants) | 8
% of lasmiditan dose | 2.91 (0.561)

8. Secondary Outcome: Renal Clearance (CLR)
Description: Renal clearance is the volume of plasma completely cleared of lasmiditan by the kidneys per unit time and calculated as CLR = Aeu/AUC0-x (where Aeu = amount of lasmiditan excreted in urine over a sampling interval; x is the last interval collected; for lasmiditan only).
Time Frame: as for outcome 6
Population: All enrolled participants who received at least one dose of the study drug and had evaluable [14C]-lasmiditan PK data.
Measure: Mean (Standard Deviation); unit: liter per hour (L/hr)
Arm/Group | [14C]-Lasmiditan
Number analyzed (Participants) | 8
liter per hour (L/hr) | 2.89 (1.12)

9. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Safety assessed from time of consent through end of study (up to 49 days). A summary of all reported serious adverse events (SAE) and other adverse events regardless of causality are provided in the Adverse Events module of this record.
Time Frame: Up to 49 days
Population: All enrolled participants who received at least one dose of the study drug and had at least 1 post-dose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | [14C]-Lasmiditan
Number analyzed (Participants) | 8
Participants
  Adverse Events (AEs) | 5
  Serious Adverse Events (SAEs) | 0

ADVERSE EVENTS:
Time Frame: Up To 49 Days
Description: All enrolled participants who received at least one dose of study drug and had at least one post-dose safety assessment.
Arm/Group | [14C]-Lasmiditan
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [14C]-Lasmiditan (N=8)
External ear pain (Ear and labyrinth disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Feeling drunk (General disorders) | 1 (1)
Post procedural contusion (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 2 (2)
Sensory disturbance (Nervous system disorders) | 1 (1)
Euphoric mood (Psychiatric disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the study and its results shall not be publicized in any form without prior consent of the Sponsor. Such approval is necessary to prevent premature disclosure of trade secrets and other confidential information.

DOCUMENTS (2):
  • Study Protocol (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT03040362/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT03040362/SAP_001.pdf